CLINICAL TRIAL: NCT07328958
Title: Effect of Titrated Administration of Ciprofol Combined With Remifentanil on Perioperative Hypotension in Elderly Patients Undergoing Laparoscopic Abdominal Surgery: A Randomized Controlled Trial
Brief Title: Effect of Titrated Administration of Ciprofol on Perioperative Hypotension in Elderly Patients Undergoing Laparoscopic Abdominal Surgery: A Randomized Controlled Trial
Acronym: TAPH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, SanQing Jin, professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025ZSLYEC-415
Record Dates: First submitted 2025-11-21; First posted 2026-01-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Hypotension During Surgery
Keywords: elderly; general anesthesia; titrated; ciprofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Data Analyst
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- controled group (No Intervention): Patients in this group will undergo anesthesia induction and maintenance with ciprofol and remifentanil. Induction will be performed with intravenous bolus administration of ciprofol at a dose of 0.4 mg/kg and remifentanil at a dose of 1-2μg/kg, followed by a neuromuscular blocker to facilitate tracheal intubation. During surgery, anesthetic doses will be adjusted at the discretion of the anesthesiologist, based on the patient's physiological parameters and surgical conditions. Depth of anesthesia will be continuously monitored; however, the monitoring results will remain blinded to the attending anesthesiologist.
- titrated group (Experimental): In this group, anesthesia induction was performed with continuous infusion of ciprofol and remifentanil until loss of consciousness (OAA/S score = 1), followed by administration of a neuromuscular blocker to facilitate tracheal intubation. After intubation, anesthesia was maintained with ciprofol (0.4-3 mg/kg/h) and remifentanil (0.01-0.5 µg/kg/min) until the end of surgery. Depth of anesthesia was adjusted intraoperatively to maintain BIS at approximately 50.
  Interventions: Drug: titrated anesthesia

INTERVENTIONS:
Drug: titrated anesthesia — Anesthesia induction and maintenance will be performed with ciprofol and remifentanil. During the entire procedure, infusion rates will be adjusted according to a target BIS value of approximately 50, with anesthetic dosing continuously modified in response to BIS monitoring. The attending anesthesiologist will titrate anesthetic delivery based on BIS guidance rather than routine clinical judgment alone.
  Arms: titrated group

SUMMARY:
Elderly patients are frequently burdened with age-associated comorbidities and frailty, accompanied by physiological changes such as vascular stiffening, cardiac dysfunction, and impaired autonomic regulation. These factors not only increase the risk of adverse perioperative outcomes but also heighten sensitivity to anesthetic agents, making elderly patients particularly susceptible to anesthesia-related complications, especially hypotension. Consequently, optimizing anesthesia strategies for this high-risk population has become a critical goal in perioperative management.

Titrated anesthesia, which individualizes anesthetic drug delivery based on patient response to achieve predefined endpoints, offers a potential approach to mitigating anesthetic risks. Ciprofol, a novel intravenous anesthetic, has been associated with less hemodynamic suppression compared with traditional agents; however, higher single doses may still predispose patients to hypotension. Remifentanil, an ultra-short-acting opioid, exerts significant cardiovascular depressive effects, further contributing to perioperative hypotension.

It is hypothesized that titrated administration of anesthetic agents during both the induction and maintenance phases, compared with conventional fixed-dose protocols, may reduce the incidence of perioperative hypotension in elderly patients.

DETAILED DESCRIPTION:
This study aims to investigate whether titrated anesthesia can provide more stable hemodynamic conditions during surgery and whether this approach is associated with improved postoperative recovery in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years, scheduled for elective laparoscopic abdominal surgery
* American Society of Anesthesiologists (ASA) physical status I-III
* Requirement for invasive arterial blood pressure monitoring

Exclusion Criteria:

* Participation in other clinical trials that may interfere with the intervention or outcomes of this study
* Severe hepatic or renal disease (GFR ≤30 mL/min/1.73 m², requirement for renal replacement therapy, or Child-Pugh class C liver function)
* Uncontrolled severe hypertension (preoperative SBP ≥180 mmHg or DBP ≥110 mmHg)
* Patients with severe mental disorders (such as schizophrenia), epilepsy, or Parkinson's disease, severe cognitive or intellectual impairment, severe visual or hearing impairments affecting assessment, or long-term alcohol abuse or use of sedative/analgesic medications;
* Known allergy to drugs used in this study
* Requirement for continuous vasopressor infusion before surgery, or intraoperative need for prolonged hemodynamic manipulation due to surgical factors
* Anticipated blood loss >15% of estimated blood volume
* Expected surgical duration <1 hours or >6 hours
* Expected postoperative hospital stay <72 hours

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-01-16 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of intraoperative hypotension. | From induction of general anesthesia to the end of surgery, assessed intraoperatively for up to 6 hours.
  Hypotension is defined as at least one episode of mean arterial pressure (MAP) <65 mmHg sustained for at least 1 minute.

SECONDARY OUTCOMES:
the time-weighted area under the curve (TWA) for MAP <65 mmHg during the anesthesia period | From induction of general anesthesia to the end of surgery, assessed intraoperatively for up to 6 hours.
  calculated as AUC / total time of anesthesia
cumulative dose of norepinephrine and the proportion of patients requiring vasoactive support; | From induction of general anesthesia to the end of surgery, assessed intraoperatively for up to 6 hours.
  the cumulative dose of norepinephrine administered intraoperatively (µg) and the proportion of patients who required any vasoactive medication (norepinephrine, dopamine, or ephedrine) during the anesthesia period.
the time-weighted area under the curve (TWA) for MAP <0.8 baseline during the anesthesia period | From induction of general anesthesia to the end of surgery, assessed intraoperatively for up to 6 hours.
  caculate as area under the curve / total anesthesia time
Time to first hypotension | From induction of general anesthesia to the end of surgery, assessed intraoperatively for up to 6 hours.
  The time to first hypotension during anesthesia
CI trend during anesthesia | From induction of general anesthesia to the end of surgery, assessed intraoperatively for up to 6 hours.
  CI data will be collected by the device and extracted for analysis.
The time periods with a higher incidence of hypotension between the two groups | From induction of general anesthesia to the end of surgery, assessed intraoperatively for up to 6 hours.
  The time is divided into four parts: induction period, post-induction period, surgical period, and early postoperative period
Total dose of ciprofol and remifentanil during surgery | From induction of general anesthesia to the end of surgery, assessed intraoperatively for up to 6 hours.
  The total doses of ciprofol and remifentanil administered per hour throughout the entire surgical procedure.
Whether blood pressure variability (CV) and the average rate of blood pressure variation (ARV) are different. | From induction of general anesthesia to the end of surgery, assessed intraoperatively for up to 6 hours.
  Both CV and ARV will be calculated using the formulas provided in the reference literature.
The incidence of severe intraoperative hypotension | From induction of general anesthesia to the end of surgery, assessed intraoperatively for up to 6 hours.
  Severe intraoperative hypotension is defined as MAP < 55 mmHg
Time from discontinuation of anesthetic drugs to awakening. | From discontinuation of anesthetic drugs to awakening, assessed up to 2 hours postoperatively.
  Awakening is defined as the first eye opening in response to a verbal command.
the rate of postoperative delirium | Postoperatively (4-6 hours), Day 1, Day 2, Day 3
  Postoperative delirium is assessed using the Chinese version of the 3D-CAM scale. The Chinese version of the 3D-CAM has a sensitivity ranging from 84.6% to 87.2% and a specificity ranging from 96.7% to 97.4%. If a patient is admitted to the ICU, the CAM-ICU scale will be used to evaluate them for delirium.
Postoperative complications | 30 days after the operation
  The evaluation of postoperative complications will be conducted using Futier's classification system for postoperative complications, with the primary basis for assessment being medical record data and follow-up data.
All-cause mortality within 30 days after surgery. | 30 days after operation
  All-cause mortality is defined as death from any cause occurring within 30 days following surgery.
Hospital readmission within 30 days after surgery | 30 days postoperatively.
  Readmission is defined as any unplanned hospital admission occurring within 30 days after surgery.
The lowest MAP during anesthesia | From induction of general anesthesia to the end of surgery, assessed intraoperatively for up to 6 hours.
  The lowest MAP during anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cannon JW. Hemorrhagic Shock. N Engl J Med. 2018 Jan 25;378(4):370-379. doi: 10.1056/NEJMra1705649. No abstract available. PMID 29365303
- [Background] Marchant A, Hartley MR. The action of pokeweed antiviral protein and ricin A-chain on mutants in the alpha-sarcin loop of Escherichia coli 23S ribosomal RNA. J Mol Biol. 1995 Dec 15;254(5):848-55. doi: 10.1006/jmbi.1995.0660. PMID 7500355
- [Background] Eisler I, Dare C, Russell GF, Szmukler G, le Grange D, Dodge E. Family and individual therapy in anorexia nervosa. A 5-year follow-up. Arch Gen Psychiatry. 1997 Nov;54(11):1025-30. doi: 10.1001/archpsyc.1997.01830230063008. PMID 9366659
- [Background] Gol'dberg VA. [The use of Difril in patients with chronic coronary insufficiency]. Klin Med (Mosk). 1968 Jun;46(6):100-3. No abstract available. Russian. PMID 5710560
- [Background] Bernasconi S, Vanelli M, Nori G, Siracusano MF, Marcellini C, Butturini A, De Luca F. Serum TSH, T4, T3, FT4, FT3, rT3, and TBG in youngsters with non-ketotic insulin-dependent diabetes mellitus. Horm Res. 1984;20(4):213-7. doi: 10.1159/000179999. PMID 6439616
- [Background] Salmasi V, Maheshwari K, Yang D, Mascha EJ, Singh A, Sessler DI, Kurz A. Relationship between Intraoperative Hypotension, Defined by Either Reduction from Baseline or Absolute Thresholds, and Acute Kidney and Myocardial Injury after Noncardiac Surgery: A Retrospective Cohort Analysis. Anesthesiology. 2017 Jan;126(1):47-65. doi: 10.1097/ALN.0000000000001432. PMID 27792044
- [Background] Maheshwari K, Turan A, Mao G, Yang D, Niazi AK, Agarwal D, Sessler DI, Kurz A. The association of hypotension during non-cardiac surgery, before and after skin incision, with postoperative acute kidney injury: a retrospective cohort analysis. Anaesthesia. 2018 Oct;73(10):1223-1228. doi: 10.1111/anae.14416. Epub 2018 Aug 24. PMID 30144029
- [Background] D'Souza AW, Hissen SL, Manabe K, Takeda R, Washio T, Coombs GB, Sanchez B, Fu Q, Shoemaker JK. Age- and sex-related differences in sympathetic vascular transduction and neurohemodynamic balance in humans. Am J Physiol Heart Circ Physiol. 2023 Oct 1;325(4):H917-H932. doi: 10.1152/ajpheart.00301.2023. Epub 2023 Aug 18. PMID 37594483
- [Background] Abdellatif M, Rainer PP, Sedej S, Kroemer G. Hallmarks of cardiovascular ageing. Nat Rev Cardiol. 2023 Nov;20(11):754-777. doi: 10.1038/s41569-023-00881-3. Epub 2023 May 16. PMID 37193857
- [Background] Brauer D. [Evaluation of medical data using statistics software: the program packet ABSTAT]. Z Arztl Fortbild (Jena). 1988;82(18):905-8. No abstract available. German. PMID 3213092